CLINICAL TRIAL: NCT05621473
Title: Comparing the Safety and Efficacy of EDUG-guided Tunnel PICC With Conventional PICC in Immunocompromised Patients: a Multicenter, Prospective, Randomized Controlled Clinical Study
Brief Title: Comparing the Safety and Effectiveness of Tunnel PICC Guided by EDUG and Conventional PICC
Acronym: PICC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong Branden Med.Device Co.,Ltd (Industry)
Collaborators: Wuhan University (Other); Enshi Clinical College of Wuhan University (Unknown); Jingzhou Central Hospital (Other); The Central Hospital of Huanggang (Other); Hubei Cancer Hospital (Other); Yichang Central People's Hospital (Other); Sinopharm Gezhouba Group Central Hospital (Unknown); Central Hospital of Xiaogan (Other); Xiaogan First People's Hospital (Unknown); Wuhan Central Hospital (Other); Xiangyang Central Hospital (Other); Xiangyang No.1 People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: brandentech-001
Record Dates: First submitted 2022-09-26; First posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: the Incidence of PICC-related Complications
MeSH Terms: interventions — Catheterization, Peripheral

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- trial group (Experimental): This arm of patients received tunnel PICC interventions
  Interventions: Device: PICC
- control group (Experimental): This arm of patients received normal PICC interventions
  Interventions: Device: PICC

INTERVENTIONS:
Device: PICC — Tunnel PICC puncture technology is a perfect combination of ultrasound-guided puncture, ECG lead technology, PICC and subcutaneous tunnel. The valve conduction PICC is equipped with an integrated ECG lead Doppler ultrasound machine. Before the catheter is placed, in the yellow area, in the ultrasound mode, evaluate the blood vessel condition, measure the blood flow velocity, and correctly select the puncture site. When the catheter is pushed close to the superior vena cava, the electrocardiograph mode is switched to complete the precise positioning of the catheter according to the principle of ECG positioning technology. A subcutaneous tunnel was prepared in the green area, and the PICC at the puncture site in the yellow area was introduced to the green area and carefully bandaged. Whole-process integrated operation, simple and efficient operation.
  Other Names: Peripherally inserted central venous catheter

SUMMARY:
This study was designed as a prospective, multicenter, randomized controlled study, with the incidence of postoperative complications as the main observation end point. It was a superiority design.The purpose of this study was to compare the incidence of complications associated with EDUG-guided subcutaneous tunneling and conventional puncture after peripheral vein placement of PICCs

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old;
* Immunocompromised patients, including:

  ① Patients with congenital T cell/B cell deficiency or macrophage disorder;

  ② Patients with solid malignant tumors or hematological malignancies;

  ③ Patients with AIDS;

  ④ Patients undergoing splenectomy or solid organ transplantation;

  ⑤ Patients with rheumatic diseases and treated with immunomodulatory drugs;
* Follow the doctor's advice to perform PICC catheterization for the first time;
* No serious cardiovascular disease, such as atrial fibrillation, pulmonary heart disease, severe conduction block, etc., before catheter placement;
* Patients who have not participated in other clinical studies;
* Patients who voluntarily participate in the clinical study and can cooperate with the clinical follow-up.

Exclusion Criteria:

* Known allergy to catheter material;
* History of infection, injury or radiation therapy at the puncture site;
* There is a history of venous thrombosis or surgical operation at the puncture site;
* Severe abnormal coagulation function;
* Superior vena cava compression syndrome;
* Radical mastectomy for breast cancer or axillary lymph node dissection on the operative side of the limb;
* Pacemaker and arteriovenous fistula ipsilateral limb.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-07-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
rate of PICC-related complications | 6 months after operation
  Observe and record the incidence of catheter-related complications during catheter placement, such as bleeding, subcutaneous congestion, lymphatic exudation, phlebitis (bacterial phlebitis, mechanical phlebitis, thrombophlebitis), infection (local infection, tunneling) Infection, catheter-related bloodstream infection), thrombosis (symptomatic thrombosis, asymptomatic thrombosis), catheter ectopic, medical adhesive-related skin injury, catheter injury and blockage, etc.

SECONDARY OUTCOMES:
time of catheter indwelling | Intraoperative (Time from successful catheter insertion to extubation)
  Time from successful catheter insertion to extubation
rate of unplanned extubation | through study completion, an average of 4months
  the incidence of unplanned extubation
success rate of one-time catheter placement | one hour
operation time | one hour
score of operation convenience | one hour
score of patient comfort | one hour

IPD SHARING:
Plan to Share IPD: No